CLINICAL TRIAL: NCT01240200
Title: Satisfaction of Treatment Among Elderly Patients With Insulin Therapy Using Pens for a Basal Insulin Treatment (STEP IT UP a BIT)
Brief Title: Satisfaction of Treatment Among Elderly Patients With Insulin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00046366
Record Dates: First submitted 2010-11-09; First posted 2010-11-15 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; elderly; insulin injections
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vial & Syringe (Period 1) / Pen (Period 2) (Active Comparator): Crossover phase: patients randomized to the sequence: Insulin glargine vial and syringe in Period 1 and Insulin glargine SoloSTAR pen in Period 2.
  Interventions: Drug: Glargine; Device: glargine via insulin pen
- Pen (Period 1) / Vial & Syringe (Period 2) (Experimental): Crossover phase: patients randomized to the sequence: Insulin glargine SoloSTAR® pen in Period 1 and Insulin glargine vial and syringe in Period 2.
  Interventions: Drug: Glargine; Device: glargine via insulin pen

INTERVENTIONS:
Drug: Glargine — oral antidiabetic agents plus once daily insulin glargine via an insulin syringe
  Other Names: Lantus
Device: glargine via insulin pen — oral antidiabetic agents plus insulin glargine in a pre-filled pen
  Other Names: Solostar

SUMMARY:
Several studies have shown that high blood sugar (glucose) levels are associated with diseases caused by diabetes. Controlling the glucose may prevent these complications. As people age, their bodies become unable to make enough insulin to control the blood sugars. Pills used to treat diabetes may help for a while, but many times this does not last. When the blood sugar is too high, insulin is frequently recommended and used to treat diabetes. Insulin is often started by adding a long-acting insulin to the medicines a patient already takes. In this study, glargine insulin will be taken together with the diabetes pills currently being used. Glargine is a long-acting insulin which is given under the skin once a day. Glargine is approved for use in the treatment of patients with diabetes by the FDA (Food and Drug Administration).

Currently, insulin delivery is only available as a shot. The purpose of this study is to compare how satisfied patients are when using two different types of insulin shots. Specifically, this study aims to determine if people over 65 years old are more satisfied taking insulin shots by pens or syringes. Everyone who joins in this study will have a chance to use the insulin syringes and the insulin pens.

The ability of patients to give themselves shots can affect how well the sugar is controlled. As people age, medical and other problems may develop that affect their ability to do certain things. Another aim of this study is to determine if the ability to use an insulin pen and insulin syringe is affected by age or some other problem.

During this study, participants will be treated with insulin given by a syringe for 12 weeks and by a pen for 12 weeks. Questionnaires will be given to determine satisfaction with treatment throughout the study. The investigators hypothesize that among elderly patients with type 2 diabetes mellitus failing oral agent therapy, treatment with basal insulin via a pen device results in higher treatment satisfaction scores and more accurate dosing than treatment with basal insulin via conventional vial and syringe methods.

A total of 56 subjects with type 2 diabetes will be recruited into this study. The site for the study is Grady Memorial Hospital clinics in Atlanta, Georgia.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥60 years
2. History of type 2 diabetes of >3 months duration
3. Current use oral antidiabetic agents and/or diet to treat the diabetes
4. A1c ≤10.0% and fasting glucose ≤300 mg/dL
5. A1c ≥7.0% and/or fasting glucose ≥150 mg/dL

Exclusion Criteria:

1. Subjects with a known allergy to glargine or any of its metabolites
2. Subjects unwilling to self-inject insulin
3. Inability to self-monitor blood glucose
4. Current or previous use of insulin for more than 6 continuous months prior to study enrollment
5. Subjects with documented clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), corticosteroid therapy, impaired renal function (creatinine >3.0 mg/dL), uncontrolled endocrine disorders associated with increased insulin resistance such as acromegaly, Cushing's syndrome, or hyperthyroidism
6. Mental condition rendering the subject unable to understand the nature, scope and/or possible consequences of the study
7. Inability or unwillingness to provide informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoper Newton, MD, Principal Investigator — Emory University SOM; Dawn Smiley, MD, MSCR, Principal Investigator — Emory University SOM
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of subjects started in January 2011 and all study participation was completed in December 2012. Patients were recruited from the Grady Memorial Hospital Diabetes Clinic in Atlanta, Georgia.
Pre-assignment Details: Of the 56 individuals who consented to take part in the study, 7 were removed prior to being randomized to a group (2 did not meet eligibility criteria and 5 withdrew consent prior to group assignment). Those who were not randomized were not considered to be enrolled in the study as group assignment was never determined.
Groups:
- Vial & Syringe (Period 1) / Pen (Period 2): Crossover study group where participants were randomized to the sequence of insulin glargine via vial and syringe in Period 1 and insulin glargine via SoloSTAR pen in Period 2.
- Pen (Period 1) / Vial & Syringe (Period 2): Crossover study group where participants were randomized to the sequence of insulin glargine via SoloSTAR® pen in Period 1 and insulin glargine via vial and syringe in Period 2.
Period: 12-week Crossover Phase - Period 1
Arm/Group | Vial & Syringe (Period 1) / Pen (Period 2) | Pen (Period 1) / Vial & Syringe (Period 2)
Started | 25 | 24
Completed | 23 | 23
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Period: 12-week Crossover Phase - Period 2
Arm/Group | Vial & Syringe (Period 1) / Pen (Period 2) | Pen (Period 1) / Vial & Syringe (Period 2)
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes the 46 participants who completed the trial (23 in Vial & Syringe to Pen group and 23 in Pen to Vial & Syringe group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Vial & Syringe (Period 1) / Pen (Period 2) | Pen (Period 1) / Vial & Syringe (Period 2) | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (5.8) | 70.6 (4.4) | 68.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Treatment Satisfaction Questionnaire: Status (DTSQs) Score
Description: Treatment satisfaction was assessed using the Diabetes Treatment Satisfaction Questionnaire: Status (DTSQs). The questionnaire contains eight items scored on a seven-point scale where 0 = very dissatisfied and 6 = very satisfied. The satisfaction score is obtained from summing responses to questions 1, 4, 5, 6, 7, and 8 and the total score can range from 0 to 36. Higher scores indicate higher satisfaction with diabetes treatment.
Time Frame: Baseline, Week 12
Population: This analysis includes participants who completed the baseline and week 12 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vial & Syringe (Period 1) / Pen (Period 2) | Pen (Period 1) / Vial & Syringe (Period 2)
Number analyzed (Participants) | 23 | 23
units on a scale
  Baseline | 28.2 (7.0) | 31.5 (4.9)
  Week 12 | 32.2 (5.2) | 34.2 (2.3)

2. Primary Outcome: Diabetes Treatment Satisfaction Questionnaire: Change (DTSQc) Score
Description: Treatment satisfaction after crossover into the second treatment period was assessed using the Diabetes Treatment Satisfaction Questionnaire: Change (DTSQc). The questionnaire contains eight items scored on a seven-point scale where -3 = much less satisfied now and 3 = much more satisfied now. The satisfaction score is obtained from summing responses to questions 1, and 4 through 8 (the remaining two items assess perceived blood sugar levels). The total score can range from -18 to 18. Higher scores indicate higher satisfaction with the new diabetes treatment, compared to prior treatment, while scores below 0 mean that satisfaction with the new delivery method of insulin in Period 2 is lower than satisfaction with the delivery method in Period 1.
Time Frame: Week 24
Population: This analysis includes participants who completed the week 12 and week 24 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vial & Syringe (Period 1) / Pen (Period 2) | Pen (Period 1) / Vial & Syringe (Period 2)
Number analyzed (Participants) | 23 | 23
units on a scale | 16.4 (2.7) | -2.3 (10.0)

3. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: Hemoglobin A1c (HbA1c) measures the average percentage of blood sugar over the past 2 to 3 months. HbA1c levels below 5.7% are considered normal. Persons with values between 5.7% and 6.4% are considered at high risk of developing diabetes while those with values of 6.5% and above are diagnosed with diabetes. HbA1c can reduce with management of diabetes through diet, exercise, and medication.
Time Frame: Baseline, Week 12
Population: Participants with HbA1c measurements at baseline and week 12 are included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of Hemoglobin A1c
Arm/Group | Vial & Syringe (Period 1) / Pen (Period 2) | Pen (Period 1) / Vial & Syringe (Period 2)
Number analyzed (Participants) | 23 | 23
percentage of Hemoglobin A1c
  Baseline | 8.7 (1.1) | 8.5 (1.3)
  Week 12 | 7.6 (0.8) | 7.6 (1.0)

4. Secondary Outcome: Fasting Blood Glucose
Description: Blood sugar levels are influenced by the size and types of food consumed during the last meal and the production and response to insulin. Fasting blood glucose levels of less than 100 milligrams per deciliter (mg/dL) are considered normal. Values between 100 and 125 mg/dL indicate prediabetes and values of 126 mg/dL and higher indicate diabetes. Fasting blood glucose levels can lower depending on food consumed and medications.
Time Frame: Baseline, Week 12
Population: Participants with fasting blood glucose measurements at baseline and week 12 are included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Pen (Period 1) / Vial & Syringe (Period 2): Crossover study group of insulin glargine via SoloSTAR® pen in Period 1 and insulin glargine via vial and syringe in Period 2.
Arm/Group | Vial & Syringe (Period 1) / Pen (Period 2) | Pen (Period 1) / Vial & Syringe (Period 2)
Number analyzed (Participants) | 23 | 23
mg/dL
  Baseline | 159 (47) | 157 (38)
  Week 12 | 126 (19) | 134 (32)

5. Secondary Outcome: Percent of Participants With Dosing Errors
Description: Percentage of participants who had dosing errors during the course of the study (both study periods). Participants were instructed on using each device and practiced preparing and injecting the insulin dose into a pillow to assess accuracy with each method of delivering insulin. Dosing errors were defined as inaccurate preparation or injection by less than or equal to 10% of the intended dose, independent of vision and dexterity function.
Time Frame: Week 24
Population: All participants completing the study are included in this analysis (23 in dosing sequence 1 and 23 in dosing sequence 2).
Measure: Number; unit: percentage of participants
Groups:
- Vial & Syringe: Participants from both dosing sequences (Period 1 and Period 2) using a vial and syringe during the study to self-administer insulin glargine.
- SoloSTAR Pen: Participants from both dosing sequences (Period 1 and Period 2) using the SoloSTAR Pen during the study to self-administer insulin glargine.
Arm/Group | Vial & Syringe | SoloSTAR Pen
Number analyzed (Participants) | 46 | 46
percentage of participants | 90 | 20

6. Secondary Outcome: Number of Hypoglycemic Events
Description: The number of hypoglycemic events occurring during the 24-week study period is reported here. For the purposes of this study, hypoglycemia is defined as a capillary and/or laboratory blood glucose value of less than 70 mg/dL.
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: hypoglycemic events
Arm/Group | Vial & Syringe | SoloSTAR Pen
Number analyzed (Participants) | 46 | 46
hypoglycemic events | 72 | 36

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time study treatment began through the completion of both 12-week periods of the study (up to 24 weeks). Twenty-five participants began the vial and syringe delivery method in Period 1 and 23 participants began this intervention in Period 2, resulting in 48 participants receiving this intervention. For the insulin pen delivery method, 24 participants began in Period 1 and 23 began in Period 2, for a total of 47 participants receiving this intervention.
Groups:
- Vial and Syringe: Participants, from both dosing sequences (Period 1 and Period 2), using a vial and syringe during the study to self-administer insulin.
- SoloSTAR Pen: Participants, from both dosing sequences (Period 1 and Period 2), using the SoloSTAR Pen during the study to self-administer insulin.
Arm/Group | Vial and Syringe | SoloSTAR Pen
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 22/48 | 15/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vial and Syringe (N=48) | SoloSTAR Pen (N=47)
Hypoglycemia (Endocrine disorders) | 22 (72) | 15 (36) — Blood glucose <70mg/dL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No